CLINICAL TRIAL: NCT07347769
Title: Study of the Serotype and Genotype of BK Virus in Kidney Transplant Recipients and Their Donors to Identify Individuals at Risk of Nephropathy
Acronym: TYPIK
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0247; 2025-A02381-48 (Other: ID RCB)
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Nephropathy; Opportunistic Viral Infection; Polyoma Virus Nephropathy; BK Nephropathy; BK Viremia; BKV DNAemia; BK Virus Infection; BK Polyomavirus; Immune Response; Neutralizing Antibodies
Keywords: TTV; BK polyomavirus; neutralizing antibodies; ELISPOT BKV; genotype; miRNA BKV; urinary chimiokine
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will retained plasma, whole blood and urine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to characterize the urinary replication of BK polyomavirus (BKV) in kidney transplant recipients. Although BKV reactivation after transplantation is well established, the origin of the replicating virus remains uncertain. Current evidence suggests that BKV detected in recipients may originate either from the transplanted kidney (donor-derived) or from viral reactivation in the recipient. The evaluation of new biomarkers to predict BKV replication are needed.

This study seeks to address the following key questions:

* Origin of the replicating virus: Is the BKV detected in the recipient identical to the virus originating from the donor kidney?
* Host immune response and viral genotype: Is there an association between the recipient's immune response and the genotype of the replicating BKV?
* Differences in immune response according to viral replication profile: Does the immune response differ between patients presenting isolated BKV viruria and those with both viruria and viremia?
* Can new biomarkers help predict BKV replication and viremia?

Patients will be grouped according to their BKV replication profile:

Group 1: patients with BKV viruria without viremia Group 2: patients with both BKV viruria and viremia Comparisons between these two groups will help identify whether different viral genotypes or immune responses are associated with systemic dissemination (viremia).

Kidney transplant recipients will be included if they present BKV viruria during their post-transplant follow-up. Additional blood samples will be collected during scheduled follow-up visits at the university hospital. These visits are part of routine clinical care, and no extra visits will be required specifically for the study.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant patients with a first positive BK virus viral load in urine. - BK virus viral load in urine > 3 log copies/mL.
* More than 3 months post-transplant and less than 2 years post-transplant.
* Men or women aged 18 years and older.
* Followed up at Grenoble Alpes University Hospital.
* Affiliated with social security or beneficiary of such a scheme.
* Patients who are not opposed to the TYPIK study.

Exclusion Criteria:

* Expected renal graft survival is < 6 months, estimated by an eGFR < 15 mL/min/1.73 m² at the time of BKPyV viruria
* Patients who object to the use of their data and/or samples for research purposes
* Subjects who are excluded from another study
* Subjects under administrative or judicial supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant patients with a first positive BK virus viral load in urine during the 2 years after the graft
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-06-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
To describe the prevalence and variability of different BKPyV genotypes and serotypes in a population of kidney transplant patients with BKPyV viruria/viremia. | up to 2 years
  The primary endpoint will be the classification by genotyping/serotyping of BKPyV obtained during the first viruria and the first viremia, performed using NGS and serotyping using a seroneutralization technique. The search for SNPs (single nucleotide polymorphisms) will also enable the subclassification of genotypes and better identification of patients at risk of BKPyV viremia and therefore BKPyV-induced nephropathy.

SECONDARY OUTCOMES:
Compare the viral genotype at the first viruria/viremia with the donor serotype and with the recipient serotype. | up to 2 years
  The donor serotype and recipient serotype will be obtained by seroneutralization (from I to IV) and the viral genotype at the first viremia and first viruria will be obtained by a complete sequencing technique (NGS).
Describe the evolution of urinary BKPyV viral load during infection and compare viruria between viruric-only and viremic patients. | up to 2 years
  The urinary viral load for BKPyV will be obtained by qPCR (R-Gene) and expressed in log IU/mL at the time of inclusion in the two groups and then up to 6 months post-inclusion.
Describe associations between urinary and blood BKPyV viral load and associated genotypes/the presence of a mismatch between the donor serotype and the recipient genotype. | up to 2 years
  Urinary viral load at inclusion and at the time of viremia (qPCR R-Gene technique in log IU/mL) and serotype mismatch obtained from serological data at the time of transplantation.
Describe the associations between the waiting time until the first viremia and the presence or absence of a serotype mismatch at the time of transplantation, the genotype at the time of the first viruria, the viral load at the time of the first viruria, | up to 2 years
  The time will be recorded in days between the first post-transplant viruria and viremia.
Compare the evolution of the anti-BKPyV T-cell functional response in patients with viruria alone and those also with viremia between inclusion and 6 months later. | up to 2 years
  Functional anti-BKPyV T cell response obtained by ELISpot and expressed in spots/350,000 PBMC evaluated at the time of the first viremia and the first viruria.
Describe the link between the functional response and the presence of viremia, the evolution of the BKPyV viral load in the blood, and the genotype. | up to 2 years
  Functional anti-BKPyV T cell response obtained by ELISpot and expressed in spots/350,000 PBMC at the time of viruria and urinary and blood viral load of BKPyV by qPCR (log IU/mL)
Compare the BKPyV genotype present in the renal biopsy at M3 with the urinary replicative genotype at inclusion and the donor serotype. | up to 2 years
  Genotyping of BKPyV in the renal biopsy at M3 and of replicative BKPyV in urine at inclusion will be provided by NGS.
  The donor serotype will be obtained by a seroneutralization technique.
Quantitatively describe the presence of BKPyV microRNAs in urine and compare the two groups (viremic and viruric alone). | up to two years
  The presence of BKPyV microRNA will be obtained by qPCR and given in copies/mL just before inclusion and during viruria
Describe the link between the quantity of BKPyV microRNAs and the replicative genotype. | up to 2 years
  BKPyV microRNA will be obtained by qPCR and given in copies/mL just before inclusion and genotyping of BKPyV in urine during the first viremia
Quantitatively describe the presence of urinary chemokines and compare the two groups (viremic and viruric alone). | up to 2 years
  The amount of chemokine obtained by ELISA will be given in µg/mL and will be obtained at all visits.
Describe the link between the quantity of B-KPyV chemokines at inclusion and the replicative genotype. | up to 2 years
  Obtaining urinary chemokine concentrations at inclusion in µg/mL and genotyping of BKPyV in urine at inclusion
Monitor the number of BKV viruria or viremia depending on the immunosuppressive treatment received. | up to 2 years
  Type of immunosuppressant and blood concentration of these at the time of viremia/viruria
Comparison of number of positive ELISpot in group with and without viremia (identify risk factor of viremia) | up to 2 years
  Occurrence of viremia in days relative to transplantation, number of spots on ELISpot during first viremia (BKPyV microRNA in copies/mL, serotyping of donor and recipient, and genotyping in recipient's urine)
Comparison of SV40 immunohistochemistry staining results and BKPyV PCR results on M3 biopsy | up to 2 years
  Estimate the proportion of concordances between SV40 positivity in immunohistochemistry and BKPyV PCR on the M3 biopsy (copies/µg DNA) (pos/pos; pos/neg; neg/neg; neg/pos)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie TRUFFOT, Principal Investigator — CHUGA
Locations (1):
- CHUGA, Grenoble, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bae H, Na DH, Chang JY, Park KH, Min JW, Ko EJ, Lee H, Yang CW, Chung BH, Oh EJ. Usefulness of BK virus-specific interferon-gamma enzyme-linked immunospot assay for predicting the outcome of BK virus infection in kidney transplant recipients. Korean J Intern Med. 2021 Jan;36(1):164-174. doi: 10.3904/kjim.2019.339. Epub 2020 Apr 3. PMID 32241081
- [Background] Demey B, Descamps V, Presne C, Helle F, Francois C, Duverlie G, Castelain S, Brochot E. BK Polyomavirus Micro-RNAs: Time Course and Clinical Relevance in Kidney Transplant Recipients. Viruses. 2021 Feb 23;13(2):351. doi: 10.3390/v13020351. PMID 33672313
- [Background] Gosert R, Rinaldo CH, Funk GA, Egli A, Ramos E, Drachenberg CB, Hirsch HH. Polyomavirus BK with rearranged noncoding control region emerge in vivo in renal transplant patients and increase viral replication and cytopathology. J Exp Med. 2008 Apr 14;205(4):841-52. doi: 10.1084/jem.20072097. Epub 2008 Mar 17. PMID 18347101
- [Background] Udomkarnjananun S, Kerr SJ, Francke MI, Avihingsanon Y, van Besouw NM, Baan CC, Hesselink DA. A systematic review and meta-analysis of enzyme-linked immunosorbent spot (ELISPOT) assay for BK polyomavirus immune response monitoring after kidney transplantation. J Clin Virol. 2021 Jul;140:104848. doi: 10.1016/j.jcv.2021.104848. Epub 2021 Apr 28. PMID 33979739
- [Background] Solis M, Velay A, Porcher R, Domingo-Calap P, Soulier E, Joly M, Meddeb M, Kack-Kack W, Moulin B, Bahram S, Stoll-Keller F, Barth H, Caillard S, Fafi-Kremer S. Neutralizing Antibody-Mediated Response and Risk of BK Virus-Associated Nephropathy. J Am Soc Nephrol. 2018 Jan;29(1):326-334. doi: 10.1681/ASN.2017050532. Epub 2017 Oct 17. PMID 29042457